CLINICAL TRIAL: NCT03816787
Title: Hemodynamic Changes During Dry Cupping Therapy on Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ting Li, Director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIRS for Cupping Therapy
Record Dates: First submitted 2019-01-20; First posted 2019-01-25 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Oxygen Metabolism; Muscle Spasticity
Keywords: Cupping Therapy; Near Infrared Spectroscopy
MeSH Terms: conditions — Muscle Spasticity | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dry cupping for patients of low back pain (Experimental): Patients will receive four consecutive dry cupping therapy application in one month.
  Interventions: Procedure: Negative pressure therapy
- dry cupping for health people (Active Comparator): Health people will receive four consecutive dry cupping therapy application in one month.
  Interventions: Procedure: Negative pressure therapy

INTERVENTIONS:
Procedure: Negative pressure therapy — Participants assigned to the treatment group will receive wet-cupping therapy 1 times per week for 4 weeks
  Other Names: Dry cupping therapy

SUMMARY:
This study aims to investigate the hemodynamic changes during dry cupping therapy (DCT) on low back pain. 50 patients with low back pain as experimental group and 50 healthy people as control group are treated by DCT. They will receive four consecutive WCT application in one month. Optical sensors were used to monitor the hemodynamic changes including oxyhemoglobin ([HbO2]), deoxy-hemoglobin ([Hb]) and the derived change in blood volume ([tHb]) in/surround the cupping sites during treatment. The investigators hope to interpret the curative effect of DCT from the perspective of modern hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had non-specific low back pains at least 12 weeks now.
* Healthy people who are interested in dry cupping therapy

Exclusion Criteria:

* Patients who have had non-specific low back pains at least 12 weeks now.
* Healthy people who are interested in dry cupping therapy

Exclusion Criteria:

* Patients who have low back pain due to specific and known etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome, cauda equinal syndrome).
* Patients who are inappropriate to the wet cupping treatment.

  * AIDS, Active Hepatitis, Tuberculosis, Syphilis
  * Patients who regularly take anticoagulants, antiplatelet drugs
  * Anemia, thrombocytopenia
  * Hemorrhagic disease like hemophilia
  * Diabetes
  * Severe cardiovascular disease
  * Kidney diseases (renal failure, chronic renal disease)
* Patients who have experiences of wet cupping treatment during last 3 months.
* Patients who have had treatment for low back pain during last 2 weeks.
* Patients who are in pregnancy or have plan to conception.
* Patients who have vertebra surgery or have plan of surgery.
* Patients who are inappropriate to join this trial judged by the radiologists or specialists.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-11-25 (Estimated); Study Completion 2021-05-29 (Estimated)

PRIMARY OUTCOMES:
Δ[HbO2] | all groups: up to 4 weeks
  the concentration changes of oxyhemoglobin (higher alternation means better curative effect)
Δ[Hb] | all groups: up to 4 weeks
  the concentration changes of deoxyhemoglobin (higher alternation means better curative effect)

SECONDARY OUTCOMES:
Δ[tHb] | all groups: up to 4 weeks
  the concentration changes of blood volume (higher alternation means better curative effect)
NRS | experimental group: up to 4 weeks
  Numeric Rating Scale for pain (lower score means better curative effect)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Significant and sustaining elevation of blood oxygen induced by Chinese cupping therapy as assessed by near-infrared spectroscopy — https://www.osapublishing.org/boe/abstract.cfm?uri=boe-8-1-223